CLINICAL TRIAL: NCT06614530
Title: Effectiveness of Chilipad in Enhancing Sleep Quality & Wellbeing
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Efforia, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13223
Record Dates: First submitted 2024-09-24; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Sleep; Wellness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Chilipad Docker Pro Interventional Arm (Experimental): Users will receive a Chilipad Docker Pro.
  Interventions: Device: Chilipad Docker Pro

INTERVENTIONS:
Device: Chilipad Docker Pro — The Chilipad Dock Pro is an advanced sleep system designed to optimize sleep by dynamically adjusting the bed's surface temperature. It consists of a mesh mattress pad and a Dock Pro control unit that circulates water through the pad, allowing users to customize the temperature between 55°F and 115°F. The system offers both single and dual control, making it ideal for individual or shared use. Equipped with AI-driven features, the Dock Pro can monitor sleep patterns and environmental factors to make real-time adjustments, ensuring optimal sleep conditions throughout the night. This intelligent temperature management system is enhanced when paired with the optional Sleepme Tracker, creating a personalized sleep experience.

SUMMARY:
This study tests the Chilipad Dock Pro Bed Cooling System and Sleep Tracker, focusing on how temperature affects sleep quality and well-being. Over a 35-day period, metrics captured by our Sleep Tracker and participant feedback will be used to evaluate sleep quality and assess well-being. Participation requires minimal time and effort - set-up, sleep, and check-in periodically to provide feedback.

DETAILED DESCRIPTION:
Sleep quality is a cornerstone of well-being, yet many struggle to achieve restful nights. Emerging research suggests that temperature regulation can play a vital role in sleep quality. The Chilipad Dock Pro Bed Cooling System promises to optimize sleep by maintaining an ideal temperature. Social media buzz and user testimonials have lauded its effectiveness, but scientific validation is limited.

The Chilipad Dock Pro is an advanced sleep system designed to optimize sleep by dynamically adjusting the bed's surface temperature. It consists of a mesh mattress pad and a Dock Pro control unit that circulates water through the pad, allowing users to customize the temperature between 55°F and 115°F. The system offers both single and dual control, making it ideal for individual or shared use. Equipped with AI-driven features, the Dock Pro can monitor sleep patterns and environmental factors to make real-time adjustments, ensuring optimal sleep conditions throughout the night. This intelligent temperature management system is enhanced when paired with the optional Sleepme Tracker, creating a personalized sleep experience.

This single-arm trial evaluates the impact of the ChiliPad Dock Pro Bed Cooling System on sleep quality and well-being. Participants act as their control, as placebos are impractical. Participants will be asked to sequentially add Chilipad functionality throughout the trial. The study will use validated scales like the PROMIS Sleep Disturbance Scale, Well-being Survey, and SF-36 to quantify the system's effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* in the United States
* recent purchaser or customer of Sleep.me

Exclusion Criteria:

* Individuals with severe insomnia
* Individuals with severe allergies or skin conditions
* Individuals with pacemakers or implanted medical devices
* Individuals with severe anxiety or stress disorders
* Pregnant individuals
* Individuals who travel across timezones frequently and/or sleep in their own bed less than 21 days in a month.
* Individuals with incontinence issues
* Individuals with severe mobility issues.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Deep Sleep as Measured by Sleep Me Sleep Tracker | Day 30
  A non-wearable sleep tracker that is placed under the mattress at heart level and automatically tracks sleep information.
REM Sleep as Measured by Sleep Me Sleep Tracker | Day 30
  A non-wearable sleep tracker that is placed under the mattress at heart level and automatically tracks sleep information.
Time to Sleep as Measured by Sleep Me Sleep Tracker | Day 30
  A non-wearable sleep tracker that is placed under the mattress at heart level and automatically tracks sleep information.
PROMIS Sleep Disturbance Scale: PROMIS-SD Score | 30 days
  The PROMIS Sleep Disturbance Scale is a validated and widely used assessment tool developed as part of the Patient-Reported Outcomes Measurement Information System (PROMIS) initiative. It is designed to measure the severity of sleep disturbances and disruptions experienced by individuals. This scale includes a range of questions that assess the frequency and impact of various sleep-related issues, such as difficulty falling asleep, nighttime awakenings, and restless sleep. Healthcare professionals and researchers rely on this scale to better understand and quantify sleep problems in patients, enabling them to tailor interventions and treatment strategies to address sleep-related concerns effectively.

SECONDARY OUTCOMES:
Wellbeing Survey: Wellbeing Survey Score | 30 Day
  The Wellbeing Survey used in this study is a validated tool designed to assess various aspects of participants' psychological well-being and quality of life. It includes a series of statements to which participants respond on a seven-point scale, measuring their level of agreement. This survey captures dimensions such as emotional and mental health, helping to track changes in well-being throughout the study.
36-Item Short Form Survey Instrument (SF-36): 36-Item Short Form Survey Instrument (SF-36) Score | 30 days
  The SF-36, or Short Form 36, is a widely used health-related quality of life questionnaire that consists of 36 questions designed to assess a person's physical and mental well-being. It measures various aspects of an individual's health, including physical functioning, role limitations due to physical and emotional problems, social functioning, mental health, energy and vitality, pain, and general health perceptions. The SF-36 provides a comprehensive overview of a person's health status and is frequently used in clinical research, healthcare assessments, and population health studies. Its versatility and ability to assess multiple dimensions of health make it a valuable tool for evaluating the impact of medical interventions and health-related interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew M Amsden, MBA, Principal Investigator — Efforia, Inc

IPD SHARING:
Plan to Share IPD: Undecided